CLINICAL TRIAL: NCT07374770
Title: The Effect of a Mindfulness-Based Eating Behavior Training on Eating Attitudes in Individuals With Orthorexic Tendencies: A Randomized Controlled Study
Brief Title: The Effect of a Mindfulness-Based Eating Behavior Training on Eating Attitudes
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, ümüş özbey yücel, Associated Prof, Amasya University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AmasyaUni2
Record Dates: First submitted 2026-01-11; First posted 2026-01-29 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Orthorexia Nervosa
Keywords: eating disorders; mindfullness
MeSH Terms: conditions — Orthorexia Nervosa; Feeding and Eating Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Education group (Experimental): Education group: Participants assigned to the education group will receive structured educational sessions related to the study topic
  Interventions: Behavioral: Mindfulness based nutrition education intervention
- Control group (No Intervention): Control group: Participants assigned to the control group will receive standard of care and will not receive the investigational intervention.

INTERVENTIONS:
Behavioral: Mindfulness based nutrition education intervention — This study will be conducted using a randomized controlled experimental design. Participants will be randomly assigned to an intervention group and a control group. Individuals in the intervention group will receive a mindfulness-based eating behavior training program delivered over a six-week period, while the control group will not receive any intervention during this time. Pre- and post-intervention assessments will be administered to both groups to evaluate changes in eating-related outcomes.
  Arms: Education group

SUMMARY:
In recent years, the increasing interest in healthy eating and access to "pure" foods has led to the widespread adoption of selective and control-oriented eating attitudes. In some individuals, this situation has contributed to an increase in tendencies toward Orthorexia Nervosa (ON), in which the pursuit of healthy eating takes on a pathological dimension. ON is characterized by perfectionism related to healthy eating, intense anxiety, cognitive rigidity, and, over time, the development of guilt, avoidance behaviors, and social restriction. The promotion of such behaviors through media and social media further hinders the recognition of ON and facilitates its hidden spread. The concept of mindfulness, which has gained prominence in recent years, aims to help individuals observe bodily sensations, emotional responses, and thoughts that arise during the eating process with a nonjudgmental awareness. In the literature, the relationship between ON and mindfulness has mostly been examined through cross-sectional studies, while intervention-based studies targeting orthorexic individuals remain limited. The aim of this study is to examine the effects of a mindfulness-based eating behavior training program developed for orthorexic individuals on eating attitudes. The study will be conducted using a randomized controlled experimental design within the framework of an original program developed with contributions from expert researchers in the fields of psychology and nutrition. The effects of the training program applied to the intervention group will be evaluated comparatively with those of the control group. Data obtained from the study will be analyzed using SPSS, RStudio, and JASP software packages. The distributional properties of the variables will be examined using visual and analytical methods. Group comparisons, changes over time, and group-by-time interaction effects will be analyzed using appropriate parametric and nonparametric statistical methods, and the level of statistical significance will be set at p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Adults with the cognitive capacity to understand the online questionnaires and the training program
* Access to the internet
* Score 30 or higher on the Düsseldorf Orthorexia Scale (DOS)

Exclusion Criteria

* Presence of any neuropsychiatric disorder
* Diagnosed eating disorder
* Current participation in a mindfulness-based intervention
* Score below 30 on the Düsseldorf Orthorexia Scale (DOS)

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-02-10 (Estimated); Primary Completion 2026-06-15 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants who completed the training program | Approximately 6-8 weeks after the initiation of the study
  Completion is defined as full participation in all components of the education program during the study period.

SECONDARY OUTCOMES:
Proportion of participants who completed the six-week training program | approximately 6-8 weeks after the initiation of the study
  Completion is defined as attendance at 100% of the scheduled education sessions during the six-week training period. The outcome will be reported as the percentage of participants who met this completion criterion.

CONTACTS AND LOCATIONS:
Locations (1):
- Amasya Uni, Amasya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No